CLINICAL TRIAL: NCT03645226
Title: Gut Microbiota Across Early Stages of Synucleinopathy: From High-risk Relatives, REM Sleep Behavior Disorder to Early Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: HMRF05162876
Record Dates: First submitted 2018-07-19; First posted 2018-08-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: REM Sleep Behavior Disorder
Keywords: Idiopathic REM sleep; Parkinson's disease; Gut microbiota; Syncleinpathy
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. Stool sample will be collected by the patients for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early PD subjects converted from iRBD: 1. Chinese aged 50 or above
  2. Being capable of giving informed consent for participation of the study
  3. PD diagnosis confirmed by neurologists according to the United Kingdom Parkinson's Disease Survey Brain Bank. Assessment tools including Unified Parkinson's Disease Rating Scale (UPDRS) and Hoehn & Yahr Staging will be used for severity grading.
  4. Onset of PD symptoms of <5 years
  5. In view of the heterogeneity of PD, we will only include those patients with RBD preceding the onset of motor symptom of PD.
  Interventions: Diagnostic Test: Colonoscopy
- iRBD subjects: 1. Age-and sex-matched with PD subjects
  2. Chinese aged 50 or above
  3. Being capable of giving informed consent for participation of the study
  4. RBD diagnosis according to the International classification of sleep disorder 3rd edition (ICSD 3rd), fulfilling both the clinical and video-polysomnography (vPSG) criteria.
  Interventions: Diagnostic Test: Colonoscopy
- First degree relatives of patients with iRBD: 1. First degree relatives of patients with iRBD;
  2. Age-and sex-matched with PD subjects
  3. Chinese aged 40 or above;
  4. Absence of dream enactment behaviors;
  5. Not cohabiting with proband
  Interventions: Diagnostic Test: Colonoscopy
- Healthy Controls: 1. Age-and sex-matched with PD subjects;
  2. Chinese aged 50 or above;
  3. Being capable of giving informed consent for participation of the study;
  4. Without a personal history or a family history of PD or RBD;
  5. Absence of dream enactment behaviors;
  6. A total score on REM Sleep Behavior Questionnaire (RBDQ-HK) less than 19, which is the suggestive cut-off of a diagnosis of RBD;
  7. Absence of RSWA as measured by v-PSG.
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Colonoscopy — All subjects will undergo standard mechanical bowel preparation with 4 liters of polyethylene glycol (Klean-Prep, Norgine Ltd., Middlesex, UK). Total colonoscopy will be performed by experienced endoscopists under conscious sedation with intravenous benzodiazepines and narcotics. A conventional intermediate-length colonoscope (Olympus Corporation, Tokyo, Japan) will be used. One mucosal biopsy will be taken in the descending colon. Biopsies will be performed using standard biopsy forces without needle (Olympus Corporation, Tokyo, Japan). Half of the samples will be immersed in 4 oC normal saline solution. All samples will be immediately sent to pathology department and will be stored in a -80 oC freeze for processing of microbiota analyses.

SUMMARY:
With the global ageing population, neurodegenerative disorders including synucleinopathy are major burdens to patients, carers and society. Synucleinopathy refers to a group of neurodegenerative diseases characterized by abnormal aggregation of alpha-synuclein protein in the central nervous system (CNS). Common examples of synucleinopathy are Parkinson's disease (PD) and dementia with Lewy bodies (DLB). Among all the premotor clinical markers that have been identified, a sleep disorder known as REM sleep behavior disorder (RBD) is associated with the highest likelihood ratio of developing PD. In addition, it has been shown that almost all RBD patients (over 80%) eventually developed neurodegenerative diseases after 14 years follow-up.

Gut microbiota and synucleinopathy In recent years, several key studies have advanced our understanding regarding the roles that brain-gut-microbiota axis plays in the pathogenesis of brain diseases, including PD. It has been shown that gut microbiota is implicated in a series of pathophysiological changes in PD, including motor deficits, microglia activation, and αSyn pathology in mice model with overexpression of αSyn. Furthermore, some microbiotas, such as enterobacteriaceae, have been shown to be positively associated with the severity of PD symptoms, including postural instability and gait difficulty.

Limitations in previous studies and knowledge gaps Nonetheless, the answers for several key questions regarding the roles of gut microbiota in the progression of synucleinopathy are still unclear. First, whether these microbiotas found in previous studies are the causes or the effects of PD. For example, medications treating PD may also affect the gut microbiome. Moreover, the microbiota may be affected by a number of factors commonly found in PD, such as constipation per se and diet. In this regard, an influential hypothesis of synucleinopahy was proposed by Braak et al at which the early premotor features including gastro-enterology symptoms, such as constipation and RBD would predate the onset of PD by some years. Thus, it is crucial to compare the microbiota among individuals at different stages of synucleinopathy. In view of slow progression of synucleinopathy and a relatively low prevalence of synucleinopathy in the general population, it is impractical to run a prospective study to examine this research question. Finally, gut microbiota is determined by both genetic and environmental factors. A family cohort design will help to understand the genetic and environmental influences on the association between microbiota and synucleinopathy.

DETAILED DESCRIPTION:
With the global ageing population, neurodegenerative disorders including synucleinopathy are major burdens to patients, carers and society. Synucleinopathy refers to a group of neurodegenerative diseases characterized by abnormal aggregation of alpha-synuclein protein in the central nervous system (CNS). Common examples of synucleinopathy are Parkinson's disease (PD), dementia with Lewy bodies (DLB) and multiple system atrophy (MSA). These diseases often run debilitating and progressive courses that affect millions of people worldwide. Up till now, there is no curable treatment and hence the development of disease-modifying agents is of utmost importance. However, it is often too late for intervention once the patients start to have the clinical presentations of these diseases. For example, it was reported that there would be at least 80% of dopaminergic neuronal loss when one starts to develop clinical motor features of PD. Thus, researchers are now focusing on identifying at-risk subjects for early intervention. There are on-going studies to look for biomarkers to identify subjects at risk for PD through population based cohort and family studies, such as the Honolulu-Asia Aging Study (HAAS) and the Prospective Validation of Risk factors for the development of Parkinson Syndromes (PRIPS). However, these studies require a very large sample size and long duration of follow-up for the outcome evaluation.1 Another approach is to follow-up subjects at preclinical or premotor phase of PD. Among all the premotor clinical markers that have been identified, REM sleep behavior disorder (RBD) is associated with the highest likelihood ratio of developing PD.2 In addition, it has been shown that almost all RBD patients (over 80%) eventually developed neurodegenerative diseases (mean follow-up years = 14.2).3 Hence, RBD helps to understand the progression of underlying neurodegenerative diseases and will serve as a potential window for neuroprotective interventions.

Gastrointestinal dysfunction and synucleinopathy In addition to RBD, gastrointestinal dysfunction often precedes the onset of motor symptoms in patients with PD. Studies reported that constipation could precede the onset of motor symptoms in PD by 20 years. Comparing to those with daily bowel open, men with bowel movement frequency of less than 1 per day had an odds ratio of 2.7 in developing PD.4 In addition, PD with co-morbid RBD seem to have more severe constipation than PD only subjects. Constipation and other gastrointestinal dysfunction are also more common in patients with iRBD than healthy controls.5 According to Braak staging, the involvement of pontine areas (Stage 2) could result in both RBD and constipation. Hence, RBD and constipation may have an interactive effect in predicting synucleinopathy.6

What is gut microbiota and its associations with PD In recent years, several key studies have advanced our understanding regarding the roles that brain-gut-microbiota axis plays in the pathogenesis of brain diseases, including PD.7 It has been shown that gut microbiota is implicated in a series of pathophysiological changes in PD, including motor deficits, microglia activation, and αSyn pathology in mice model with overexpression of αSyn.8 Furthermore, some microbiotas, such as enterobacteriaceae, have been shown to be positively associated with the severity of PD symptoms, including postural instability and gait difficulty.9 The crucial roles of gut microbiota in the pathogenesis of PD are also evidenced by other observations.10 For example, catecholamine levels are altered in germ-free mice when compared with control mice. Antibiotics are able to reduce Firmicutes/Bacteroidetes ratio and prevent nigrostriatal dopaminergic neurodegeneration in MPTP model of PD. Probiotics increase production of L-DOPA by Bacillus and alleviate constipation in PD patients. Fecal transplantation decreased GI pathology in neurodegenerative diseases. Finally, H. pylori infection seems to increase symptom severity of PD. Taken together, growing evidence suggests that gut microbiota may play a critical role in pathogenesis, disease progression, and symptom fluctuation of synucleinopathy.

The exact mechanisms underlying the association between microbiota and Parkinson's disease remain unclear. It is believed that local and systemic inflammation and oxidative stress play a critical role in the pathogenesis of Parkinson's disease.11 In human subjects, it has been shown that proinflammatory dysbiosis is present in PD patients, which may trigger inflammation-induced misfolding of α-Syn and development of PD pathology.12 Gut microbiota is considered as an important but neglected organ for immune and inflammation. It has been shown that anti-inflammatory butyrate-producing bacteria and proinflammatory proteobacteria were significantly more abundant in feces and mucosa samples in patients with PD than healthy controls.12 Taken together, these findings suggest that gut microbiota, which is likely to increase inflammatory pathway, plays a critical role in the pathogenesis of Parkinson's disease.

Limitations and knowledge gaps Nonetheless, the answers for several key questions regarding the roles of gut microbiota in the progression of synucleinopathy are still unclear. First, whether these microbiotas found in previous studies are the causes or the effects of PD should be further clarified. It has been shown that medications treating PD also affect the gut microbiome.13 Moreover, the microbiota may be affected by a number of factors commonly found in PD, such as constipation per se and diet.14. In this regard, it is crucial to compare the microbiota among individuals at different stages of synucleinopathy. In view of slow progression of synucleinopathy and a relatively low prevalence of synucleinopathy in the general population, it is impractical to run a prospective study to examine this research question. In this regard, a case-control study with high-risk subjects is able to recruit sufficient cases at different stages of synucleinopathy.

Aims:

1. To identify the differences in colonic bacterial composition in mucosa and feces among early PD converted from iRBD, iRBD, first degree relatives (FDRs) of patients with iRBD, and healthy controls;
2. To correlate the abundance of those microbiota with clinical biomarkers of synucleinopathy.

We hypothesize that

1. Colonic bacterial composition, especially those related to inflammation (such as Blautia, Coprococcus, and Roseburia), in mucosa and feces is more abundant in different stages of synucleinopathy, namely early PD without dementia (converted from iRBD), iRBD, FDRs of patients with iRBD, and healthy controls with a dose-response pattern.
2. The abundance of microbiota is associated with other biomarkers, for example, subtle motor signs and constipation, in relation to PD and RBD.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the groups criteria

Exclusion Criteria:

1. Presence of narcolepsy and other neurodegenerative diseases (except for PD group) that may give rise to RBD and RWSA;
2. A total score of the MOCA ≤ 22 and the CDR ≥ 1, indicating dementia;
3. The use of probiotics or antibiotics within three months prior to sample collection;
4. Pre-existing gastrointestinal diseases, such as inflammatory bowel disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the case-control study, we will recruit 7 groups of subjects, which represent different stages of Parkinson's disease, namely patients with PD (Braak's stages 3 or 4) without dementia, patients with iRBD (Braak's stage 2), first degree relatives of iRBD patients (Braak's stage 0 or 1), healthy controls (Braak's stage 0). In the familial study, another 3 groups of subjects will be recruited to understand the genetic and environmental influences on differential microbiotas, including spouses of iRBD, spouses of healthy controls and first degree relatives of healthy controls.
  We will document the cohabiting status and contact frequency among family members within the same family and excluded FDRs who are cohabiting with the proband or spouses who are not cohabiting with the proband. In addition, we will also recruit FDRs and spouses with and without biomarkers of neurodegeneration (such as constipation).
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Differential abundances of colonic mucosal and fecal microbial taxa by 16S ribosomal RNA sequencing across early stages of synucleinopathy | 12 months
  To investigate differential abundances of colonic mucosal and fecal microbial taxa by 16S ribosomal RNA sequencing across early stages of synucleinopathy compared with healthy controls
Abundances of fecal microbial taxa by 16S ribosomal RNA sequencing in control and iRBD families | 12 months
  To investigate the abundances of fecal microbial taxa by 16S ribosomal RNA sequencing among probands, first-degree relatives and spouses in both healthy control and iRBD families
Biomarkers of Parkinson's disease during early stages of synucleinopathy according to questionnaire and clinical interview | 12 months
  To investigate the background risk and prodromal markers according to the MDS research criteria for prodromal Parkinson's disease in each group by questionnaire and clinical interview, for example , subtle motor signs , constipation and olfactory function

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Hong Kong
  - Shatin Hospital, Shatin

IPD SHARING:
Plan to Share IPD: Undecided
In this stage, we didn't decide whcih information of IPD will share with other researchers.